CLINICAL TRIAL: NCT02180178
Title: Mainzer IntraCoronAry daTabase (MICAT). Das Coronary Slow Flow- Syndrom Und Koronare Mikrozirkulationsstörungen- Register.
Brief Title: Mainz Intracoronary Database. The Coronary Slow-flow and Microvascular Diseases Registry
Acronym: MICAT
Status: Recruiting | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Tommaso Gori, Prof., Johannes Gutenberg University Mainz
Other Study IDs: MICAT
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease; Microvascular Dysfunction
Keywords: microvascular disease; coronary artery disease; Coronary artery disease, with or without microvascular dysfuntion
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — serum samples from patients with slow flow
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Consecutive patients undergoing coronary angiography: Consecutive patients undergoing coronary angiography at the University Medical Center Mainz - no inclusion criteria specified. The absorb substudy will include consecutive patients who received an Absorb scaffold based on clinical indication.
  Interventions: Other: observational only- no intervention

INTERVENTIONS:
Other: observational only- no intervention

SUMMARY:
Primary goal of the registry is to collect prospective data on patients undergoing coronary angiography in Mainz. Following amendment of the procol, this study will also include patients who received an Aborb bioresorbable scaffold for the therapy of de novo stenoses.

DETAILED DESCRIPTION:
Patients included in the registry will be contacted by telephone at 3,6,9, 12 months and 2, 5, 10 years after the procedure. In case coronary slow flow is shown at the index procedure, 39ml of blood will be drawn for further studies.

According to the regulations of the Province Rheinland-Pfalz, national law, and with the approval of the Ethic commission of the Landesärztekammer Rheinland Pfalz, patients (n=1000) will also be retrospectively entered in the database in an anonymous way. For these patients, no specific study procedure is foreseen and the MICAT database will be only used as a platform (database of anonymous data collected during routine clinical practice).

ELIGIBILITY:
Inclusion Criteria:

* clinical indication to coronary angiography

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with clinical indication for coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-09; Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | baseline to 10 years
  Incidence of major adverse events (death, death of cardiac cause, TLR - target lesion revascularization, MI)

SECONDARY OUTCOMES:
Individual endpoints | baseline to 10 years
  Each individual endpoint of the MACE previously described
Other cardiovascular endpoints | baseline to 10 years
  TVR - target vessel revascularization, re-hospitalization, change in medications.

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Gori, PhD Dott Med e Chirurgia, Principal Investigator — University Medical Center Mainz
Locations (1):
- University Medical Center Mainz - 2 Medizinische Klinik, Mainz, Germany

REFERENCES:
- [Derived] Gori T, Weissner M, Gonner S, Wendling F, Ullrich H, Ellis S, Anadol R, Polimeni A, Munzel T. Characteristics, Predictors, and Mechanisms of Thrombosis in Coronary Bioresorbable Scaffolds: Differences Between Early and Late Events. JACC Cardiovasc Interv. 2017 Dec 11;10(23):2363-2371. doi: 10.1016/j.jcin.2017.08.020. PMID 29216999
- [Derived] Puricel S, Cuculi F, Weissner M, Schmermund A, Jamshidi P, Nyffenegger T, Binder H, Eggebrecht H, Munzel T, Cook S, Gori T. Bioresorbable Coronary Scaffold Thrombosis: Multicenter Comprehensive Analysis of Clinical Presentation, Mechanisms, and Predictors. J Am Coll Cardiol. 2016 Mar 1;67(8):921-931. doi: 10.1016/j.jacc.2015.12.019. PMID 26916481